CLINICAL TRIAL: NCT05959486
Title: An Open-label, Randomized, Fasting, Single-dose, 2-sequence, 4-period, Full Replicated Crossover Study to Evaluate the Pharmacokinetics and Safety Between Single Administration of "BR6002" and Coadministration of "BR6002A" and "BR6002B" in Healthy Adult Volunteers
Brief Title: A Study to Evaluate the Pharmacokinetics and Safety Between Single Administration of "BR6002" and Coadministration of "BR6002A" and "BR6002B" Under Fasting Conditions in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: BR-ARC-CT-102
Record Dates: First submitted 2023-07-17; First posted 2023-07-25 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Gastric or Duodenal Ulcers
MeSH Terms: conditions — Duodenal Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BR6002A+BR6002B (Active Comparator)
  Interventions: Drug: BR6002A; Drug: BR6002B
- BR6002 (Experimental)
  Interventions: Drug: BR6002

INTERVENTIONS:
Drug: BR6002A — One tablet administered alone
  Arms: BR6002A+BR6002B
Drug: BR6002B — One tablet administered alone
  Arms: BR6002A+BR6002B
Drug: BR6002 — One capsule administered alone
  Arms: BR6002

SUMMARY:
The purpose of this clinical trial is to evaluate the pharmacokinetics and safety between single administration of "BR6002" and coadministration of "BR6002A" and "BR6002B" under fasting conditions in healthy adult volunteers

ELIGIBILITY:
Inclusion Criteria:

* Those who weigh 55 kg or more for men and 50 kg or more for women and have body mass index (BMI) within the range of 18.0 to 30.0kg/m2 at screening visit.
* Those who agree to rule out the possibility of their and their spouses' or sexual partners' pregnancy by using methods of contraception (In the case of a female subject, hormone drugs is excluded) accepted in clinical trial from the date of the first administration of the investigational products to 7 days after the last administration and disagrees to provide their sperm or ovum.

  *Methods of contraception accepted in clinical trial: Combined use of intrauterine device, vasectomy, tubal ligation, and barrier methods (male condom, female condom, cervical cap, diaphragm, sponge, etc.) or combined use of two or more barrier methods if spermicide is used.
* Those who sign written consent spontaneously after listening to and understanding sufficient explanation of the purpose and contents of this clinical trial, characteristics of the Investigational products, expected adverse events, etc.

Exclusion Criteria:

* Those who have clinically significant diseases or past history of the gastrointestinal system, cardiovascular system, endocrine system, respiratory system, hemato-oncologic disease, infectious disease, kidney

  & genitourinary system, neuropsychiatric system, musculoskeletal system, immune system, ENT system, skin system, ophthalmic system.
* Those who have a medical history of gastrointestinal surgery (Except for simple appendectomy, hernia surgery) or gastrointestinal diseases that may affect the absorption of drugs.
* Those who have taken drugs that induce and inhibit metabolizing enzymes such as barbiturate within 1 month prior to the first day of administration or have taken ETC, OTC, herbal medicine and health functional foods concerned about affecting this clinical trial within 10 days prior to the first day of administration. (however, participation is possible considering pharmacokinetics and pharmacodynamics such as Interaction of investigational products, half-life of concomitant drugs)
* Those who have participated in other clinical trials or bioequivalence tests and administered their investigational products within 6 months prior to the first administration date.
* In the case of a female subject, those suspected pregnancy, pregnant woman, lactating woman.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-07-14 (Actual); Primary Completion 2023-08-24 (Actual); Study Completion 2023-08-24 (Actual)

PRIMARY OUTCOMES:
AUCτ | 0-12 hours after administration
  Area under the concentration-time curve from time zero to time τ
Cmax | 0-12 hours after administration
  Maximum concentration of drug in plasma

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Center, H PLUS Yangji Hospital, Seoul, Gwanakgu, South Korea

IPD SHARING:
Plan to Share IPD: No